CLINICAL TRIAL: NCT02000492
Title: Intense School Based Physical Activity - Physiological, Cognitive and Sociological Aspects
Brief Title: Frequent Ballgames Training for 9-11 Year Old Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Claus Malta Nielsen, Municipal doktor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-3-2013-038; 18172 (Other: Styrelsen for Forskning og Innovation)
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Body Composition; Echocardiography
MeSH Terms: interventions — Running; Circuit-Based Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Football, circuit training or running 5x12 minutes or 3x 40 minutes
  Interventions: Behavioral: Football; Behavioral: Running; Behavioral: Circuit training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Football
  Arms: Training
Behavioral: Running
  Arms: Training
Behavioral: Circuit training
  Arms: Training

SUMMARY:
Inactivity among schoolchildren is a challenge to public health and for the municipality in particular. This study´s aim is to evaluate the cognitive and physical as well as social and fitness adaptations, and learning outcomes of short- and long term ball training for 9-11 years old girls and boys, and to determine to what extend the organisation (5x12 minutes og 3x40 minute a week) and type of training (ball games, circuit training or running) influence the magnitude of response.

ELIGIBILITY:
Inclusion Criteria:

* 9-11 years old girls and boys in 3rd grade in schools in Frederikssund and Copenhagen

Exclusion Criteria:

* Children with severe mental or physical disabilities

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 423 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cardiac function | 1 year
  echocardiography
Body composition | 1 year
  dual energy x-ray absorptiometry (DXA-scanning)

SECONDARY OUTCOMES:
Cognitive effect | 1 year
  computer based tests for cognitive and learning effects

OTHER OUTCOMES:
Social effects | 1 Year
  focus group Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Peter Krustrup, Professor, Principal Investigator — Centre of team sports and health, University of Copenhagen; Peter R Hansen, dr Msc, Principal Investigator — University hospital og Gentofte
Locations (1):
- Municipality of Frederikssund, Frederikssund, Denmark, Denmark

REFERENCES:
- [Derived] Larsen MN, Madsen M, Nielsen CM, Manniche V, Hansen L, Bangsbo J, Krustrup P, Hansen PR. Cardiovascular adaptations after 10 months of daily 12-min bouts of intense school-based physical training for 8-10-year-old children. Prog Cardiovasc Dis. 2020 Nov-Dec;63(6):813-817. doi: 10.1016/j.pcad.2020.05.011. Epub 2020 Jun 1. PMID 32497586
- [Derived] Larsen MN, Nielsen CM, Helge EW, Madsen M, Manniche V, Hansen L, Hansen PR, Bangsbo J, Krustrup P. Positive effects on bone mineralisation and muscular fitness after 10 months of intense school-based physical training for children aged 8-10 years: the FIT FIRST randomised controlled trial. Br J Sports Med. 2018 Feb;52(4):254-260. doi: 10.1136/bjsports-2016-096219. Epub 2016 Jun 13. PMID 27297443